CLINICAL TRIAL: NCT03008421
Title: Oral Probiotics to Reduce Vaginal Group B Streptococcal Colonization in Late Pregnancy: A Randomized Placebo-controlled Double-blinded Trial
Brief Title: Oral Probiotics to Reduce Vaginal Group B Streptococcal Colonization in Late Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alex Farr, MD PhD, Assistant Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1001-2017
Record Dates: First submitted 2016-12-27; First posted 2017-01-02 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-02

CONDITIONS: Vaginal Infection; Pregnancy Complications; Neonatal Sepsis; GBS
MeSH Terms: conditions — Vaginitis; Pregnancy Complications; Neonatal Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (GBS positive w/o infection) (Experimental): Treatment with study medication twice daily for 2 weeks (from study visit 1 to study visit 2)
  Interventions: Dietary Supplement: Astarte® (HSO Health Care GmbH, Vienna, Austria)
- Placebo group (GBS positive w/o infection) (Placebo Comparator): Treatment with placebo twice daily for 2 weeks (from study visit 1 to study visit 2)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Astarte® (HSO Health Care GmbH, Vienna, Austria) — oral intake of Astarte® (HSO Health Care GmbH, Vienna, Austria) as described
  Arms: Study group (GBS positive w/o infection)
Other: Placebo — Identical-looking oral potato-maltodextrin-based placebo
  Arms: Placebo group (GBS positive w/o infection)

SUMMARY:
In the present study, the investigators aim to evaluate the potential of oral probiotics, containing Lactobacillus strains, to eradicate and reduce the vaginal colonization with group B Streptococcus (GBS) during pregnancy. This could help to prevent neonatal morbidity and mortality by reducing the risk for neonatal sepsis, pneumonia, and meningitis, known as early-onset or late-onset GBS infection.

DETAILED DESCRIPTION:
The group B Streptococcus (GBS) or Streptococcus agalactiae is a gram-positive bacterium that is present in 10-30% of the healthy female population (1). Throughout pregnancy and the intrapartum period, maternal colonization with GBS can lead to the vertical transmission of the bacterium to the infant. This can result in neonatal sepsis, pneumonia, and meningitis, known as early-onset GBS infection, as well as in maternal urinary tract infections, arthritis, and pneumonia (2). Various strategies were tested to prevent the GBS infection. The antenatal GBS screening was successfully proven to identify colonized women, who should receive the intrapartum antimicrobial prophylaxis. This strategy led to a substantial reduction of the incidence of neonatal sepsis of almost 80% (3). As a result, the general use of a GBS screening was then integrated in the US-American recommendations, since the screening was superior to the risk-related procedure, when comparing the rates of early-onset neonatal sepsis (4). Later on, the GBS screening also became part of the recommendations of a European Consensus Conference (3).

The urogenital microflora of a healthy woman comprises approximately 50 species of organisms, which differ in composition according to the exposure to several factors. The flora of pregnant women is dominated by a variety of Lactobacillus species, which play an essential role in protecting them from genital infections (5). A deficiency in lactobacilli can upset the microbial balance in the vagina, which may result in an increased susceptibility for the colonization with pathogens such as GBS (6). As demonstrated by Gardnerella vaginalis, Lactobacillus strains can disrupt the biofilm of these pathogens in the in-vitro setting, which inhibits their growth (7). This led to the use of probiotics to populate the vagina with, in order to prevent or treat infections. The supplementation of probiotics that contain Lactobacillus strains has later been proven to improve cure rates and prevent recurrent infections (8).

At our Department, pregnancy care includes a prenatal consultation, where women register for a planned delivery between 10 + 0 (10 weeks plus 0 days) and 16 + 0 (16 weeks plus 0 days) gestational weeks. During this consultation, they undergo routine screening for asymptomatic vaginal infections by the Gram-stained analysis of their vaginal flora (9). In case of a vaginal infection, they undergo follow-up smears after 4-6 weeks. Routine pregnancy care is performed at outpatient gynecologists' offices, following the Austrian government's welfare program, documented in the official mother-child booklet. This national pregnancy care program is used for the health precautions of women and their fetuses including obligatory examinations at predetermined points (10). European guidelines recommend the antenatal screening for the vaginal colonization with group B Streptococcus (GBS) between 35 + 0 and 37 + 0 gestational weeks, which is performed on demand by the outpatient gynecologists, but not routinely covered by social health insurance in Austria (3).

During the routine registration for delivery at our Department, women will be asked to participate in our study. Assessment for eligibility will be performed in women with a (i) singleton pregnancy, (ii) without imminent miscarriage, (iii) without having recently undergone antibiotic or probiotic treatment. After informed consent, study participants will be asked to present between 34 + 0 and 36 + 0 gestational weeks for their first study visit. At this visit, a CDC-recommended combined vaginal-to-rectal swab will be taken from the introitus vaginae and anorectum. The combined incubation is known to increase the detection rate of GBS by up to 30% (11). Sterile swabs will be obtained after vaginal fluid collection from the lateral vaginal wall and posterior fornix vaginae, followed by the insertion into the anal sphincter. For the culture based method, they will be applied to a transport medium and subsequently inoculated in the microbiological laboratory. After inoculation, a selective enrichment broth will be used (TransVag Broth), followed by the incubation for 18 to 24 hours. That will be followed by a subculture using selective media for another 18 to 24 hours. If colonies are present, they will undergo extraction to determine if Group A or B streptococcus is present (12, 13). The threshold for GBS positive results will be considered as greater than 102 colony-forming units (CFU) per swab.

In case of a negative GBS screening result, women will be excluded from the study. In case of a positive GBS screening result, women will be randomized to the verum or the placebo group. The study will follow a prospective randomized placebo-controlled double-blinded mono-centric design. Randomization will be performed using Randomizer® (Institute for Medical Informatics, Statistics and Documentation, Medical University of Graz), which is a web-based patient randomization service for clinical trials. Women who are assigned to the verum group will receive a patented dietary supplement of four viable lactobacilli strains (HSO Health Care GmbH, Vienna, Austria), containing Lactobacillus crispatus Lbv88, Lactobacillus rhamnosus Lbv96, Lactobacillus jensenii Lbv116, and Lactobacillus gasseri Lbv150. This supplementation was proven to transmigrate from the intestinal lumen into the vaginal area, acting in the microbial ecosystem through a barrier effect against pathogenic microorganisms, so that symptoms related to dysbiosis and recurrent infections can be relieved or even prevented (14-16). Supplementation will include twice daily (morning/evening) oral intake for 14 days. Women in the placebo group will receive an identical-looking oral potato-maltodextrin-based placebo, which will also be given twice daily (morning/evening) for 14 days. Patients, investigators, and microbiological staff will be blinded to the treatment assignment. The composition of the study medication is as follows: L.crispatus Lbv88 (DSM 22566) 1 x 10^9 Guaranteed viable cell count (CFU/dose), L. rhamnosus Lbv96 (DSM 22560) 1 x 10^9 CFU/dose, L. jensenii Lbv116 (DSM 22567) 0.2 x 10^9 CFU/dose, L. gasseri Lbv150N (DSM 22583) 0.3 x 10^9 CFU/dose, Potato maltodextrin, Insoluble dietary fibre, and Silicium dioxide.

From each participant, a consecutive vaginal swab will be taken during the second study visit between 36 + 0 and 38 + 0 gestational weeks (i.e., 2 weeks after the first study visit). Sterile swabs will be obtained and inoculated as previously described. In case of a positive GBS screening result, (i) patients will be subsequently informed, and the result will be documented in (ii) the mother-child booklet and (iii) the PIA Fetal Database, version 5.6.16.917 (General Electric Company, GE Viewpoint, Munich, Germany). This procedure is necessary to ensure intrapartum penicillin treatment, which will follow current guidelines and routine practice (2). During both study visits, a vaginal swab will also be taken to perform Gram-stained analysis of the vaginal flora, in order to exclude women with acute infections (i.e., bacterial vaginosis, trichomoniasis, candidiasis) at study visit 1, and to gain further information on their flora.

The primary endpoint of our study will be the recovery to the GBS negative state. Secondary endpoints will include (i) the rate of early-onset neonatal sepsis (postnatal age less than 7 days), (ii) the rate of late-onset neonatal sepsis (postnatal age at more than 7 days), (iii) the gestational age at delivery, recorded as term delivery at or after 37 + 0 gestational weeks, (iv) the rate of preterm delivery, defined as delivery at or before 36 + 6 gestational weeks, (v) neonatal birthweight, defined as a the weight at the time of delivery, (vi) the rate of live birth, defined as the term or preterm delivery of an infant that had an Apgar score at 1 minute of > 0, and (vii) the mode of delivery (i.e., spontaneous vaginal birth, cesarean section, or instrumental vaginal delivery).

Per day, approximately 10 patients undergo routine registration for delivery at our department. All of them will be assessed for eligibility for the study. Approximately 60% of these patients will present with a normal vaginal flora without infection, which would lead to the number of 6/10 potentially eligible patients per day. A systematic review on the prevalence of maternal GBS colonization in Europe reported rates ranging from 6.5% to 36%. The carriage rates varied with Eastern Europe 19.7% to 29.3%, Western Europe 11% to 21%, Scandinavia 24.3% to 36%, and Southern Europe 6.5% to 32% (17). The investigators therefore conclude that the GBS colonization rates within our obstetric population will be approximately 25%. This will lead to the number of 1.5/6 potentially eligible patients per day, who could then be assigned to randomization.

The power for the present study was calculated using the dichotomized endpoint: recovery y/n. (i.e., defined as GBS negative). For the sample size calculation, the investigators assume that 43% of the women in the verum group will achieve the primary endpoint (i.e., recovery to the GBS negative state). This calculation is based on previously published clinical and preclinical data (18-20). The investigators expect a 18% recovery rate in the placebo group. Under these assumptions, the Chi-Squared test at two-sided significance level α = 0.05 will have 90% power to detect the group difference in a sample of N = 70 per group. With regard to a drop-out rate of 10%, the investigators will therefore need to screen N = 1040 at study visit 1, which would lead to 624/1040 (60%) patients without infection, of which 156/624 (25%) will be GBS-positive. Out of these, N = 78 per group will then be randomized, which would lead to N = 70 per group after the estimated drop-out of 10%. The investigators will need between 9-12 months to screen 1040 patients for study inclusion.

--

References:

1. Verani JR, McGee L, Schrag SJ, Division of Bacterial Diseases NCfI, Respiratory Diseases CfDC, Prevention. Prevention of perinatal group B streptococcal disease--revised guidelines from CDC, 2010. MMWR Recommendations and reports : Morbidity and mortality weekly report Recommendations and reports. 2010 Nov 19;59(RR-10):1-36. PubMed PMID: 21088663.
2. Ohlsson A, Shah VS. Intrapartum antibiotics for known maternal Group B streptococcal colonization. The Cochrane database of systematic reviews. 2014 Jun 10(6):CD007467. PubMed PMID: 24915629.
3. Di Renzo GC, Melin P, Berardi A, Blennow M, Carbonell-Estrany X, Donzelli GP, et al. Intrapartum GBS screening and antibiotic prophylaxis: a European consensus conference. The journal of maternal-fetal & neonatal medicine : the official journal of the European Association of Perinatal Medicine, the Federation of Asia and Oceania Perinatal Societies, the International Society of Perinatal Obstet. 2015 May;28(7):766-82. PubMed PMID: 25162923.
4. Schrag SJ, Zell ER, Lynfield R, Roome A, Arnold KE, Craig AS, et al. A population-based comparison of strategies to prevent early-onset group B streptococcal disease in neonates. The New England journal of medicine. 2002 Jul 25;347(4):233-9. PubMed PMID: 12140298.
5. Spiegel CA, Amsel R, Eschenbach D, Schoenknecht F, Holmes KK. Anaerobic bacteria in nonspecific vaginitis. The New England journal of medicine. 1980 Sep 11;303(11):601-7. PubMed PMID: 6967562.
6. Forsum U, Holst E, Larsson PG, Vasquez A, Jakobsson T, Mattsby-Baltzer I. Bacterial vaginosis--a microbiological and immunological enigma. APMIS : acta pathologica, microbiologica, et immunologica Scandinavica. 2005 Feb;113(2):81-90. PubMed PMID: 15723682.
7. Saunders S, Bocking A, Challis J, Reid G. Effect of Lactobacillus challenge on Gardnerella vaginalis biofilms. Colloids and surfaces B, Biointerfaces. 2007 Apr 01;55(2):138-42. PubMed PMID: 17234391.
8. Rayes N, Seehofer D, Hansen S, Boucsein K, Muller AR, Serke S, et al. Early enteral supply of lactobacillus and fiber versus selective bowel decontamination: a controlled trial in liver transplant recipients. Transplantation. 2002 Jul 15;74(1):123-7. PubMed PMID: 12134110.
9. Farr A, Kiss H, Hagmann M, Marschalek J, Husslein P, Petricevic L. Routine Use of an Antenatal Infection Screen-and-Treat Program to Prevent Preterm Birth: Long-Term Experience at a Tertiary Referral Center. Birth. 2015 Jun;42(2):173-80. PubMed PMID: 25677078.
10. Sperno R, Rudelstorfer R, Gruber W. [Effect of prenatal care in general practice and in the clinic on the course of pregnancy and labor]. Wiener medizinische Wochenschrift. 1985 Feb 15;135(3):65-9. PubMed PMID: 3984353. Einfluss der pranatalen Betreuung in Praxis und Klinik auf den Schwangerschafts- und Geburtsverlauf.
11. American College of O, Gynecologists Committee on Obstetric P. ACOG Committee Opinion No. 485: Prevention of early-onset group B streptococcal disease in newborns. Obstetrics and gynecology. 2011 Apr;117(4):1019-27. PubMed PMID: 21422882.
12. Baker CJ, Clark DJ, Barrett FF. Selective broth medium for isolation of group B streptococci. Applied microbiology. 1973 Dec;26(6):884-5. PubMed PMID: 4588195. Pubmed Central PMCID: 379927.
13. Larsen JW, Sever JL. Group B Streptococcus and pregnancy: a review. American journal of obstetrics and gynecology. 2008 Apr;198(4):440-8; discussion 8-50. PubMed PMID: 18201679.
14. Kiss H, Kogler B, Petricevic L, Sauerzapf I, Klayraung S, Domig K, et al. Vaginal Lactobacillus microbiota of healthy women in the late first trimester of pregnancy. BJOG : an international journal of obstetrics and gynaecology. 2007 Nov;114(11):1402-7. PubMed PMID: 17877778.
15. Kaufmann U, Domig KJ, Lippitsch CI, Kraler M, Marschalek J, Kneifel W, et al. Ability of an orally administered lactobacilli preparation to improve the quality of the neovaginal microflora in male to female transsexual women. European journal of obstetrics, gynecology, and reproductive biology. 2014 Jan;172:102-5. PubMed PMID: 24239295.
16. Domig KJ, Kiss H, Petricevic L, Viernstein H, Unger F, Kneifel W. Strategies for the evaluation and selection of potential vaginal probiotics from human sources: an exemplary study. Beneficial microbes. 2014 Sep;5(3):263-72. PubMed PMID: 24675230.
17. Barcaite E, Bartusevicius A, Tameliene R, Kliucinskas M, Maleckiene L, Nadisauskiene R. Prevalence of maternal group B streptococcal colonisation in European countries. Acta obstetricia et gynecologica Scandinavica. 2008;87(3):260-71. PubMed PMID: 18307064.
18. Ho M, Chang YY, Chang WC, Lin HC, Wang MH, Lin WC, et al. Oral Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 to reduce Group B Streptococcus colonization in pregnant women: A randomized controlled trial. Taiwanese journal of obstetrics & gynecology. 2016 Aug;55(4):515-8. PubMed PMID: 27590374.
19. De Gregorio PR, Juarez Tomas MS, Leccese Terraf MC, Nader-Macias ME. Preventive effect of Lactobacillus reuteri CRL1324 on Group B Streptococcus vaginal colonization in an experimental mouse model. Journal of applied microbiology. 2015 Apr;118(4):1034-47. PubMed PMID: 25786121.
20. Reid JN, Bisanz JE, Monachese M, Burton JP, Reid G. The rationale for probiotics improving reproductive health and pregnancy outcome. American journal of reproductive immunology. 2013 Jun;69(6):558-66. PubMed PMID: 23414386.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women btw. 34 + 0 and 36 + 0 gestational weeks
* GBS positive at GBS screening (study visit 1)
* No current vaginal infection (i.e., Nugent score 0-6 w/o other pathogens at study visit 1)

Exclusion Criteria:

* Multiple pregnancy
* Vaginal bleeding
* Current vaginal infection (i.e., bacterial vaginosis, chlamydia, trichomoniasis, candidiasis or others)
* Antibiotics < 4 weeks to randomization
* Probiotics < 4 weeks to randomization

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1058 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
GBS status | 2 weeks
  Eradication of vaginal colonization with group B Streptococcus (GBS) at study visit 2

SECONDARY OUTCOMES:
Neonatal sepsis | < 7d vs. >= 7 days post partum (early vs. late-onset)
  Rate of early-onset and/or late-onset neonatal sepsis
Gestational age at delivery | 6 weeks
  Term delivery at or after 37 + 0 gestational weeks vs. preterm delivery at or before 36 + 6 gestational weeks
Neonatal birthweight | 6 weeks
  Birthweight of the neonate at delivery
Live birth | 6 weeks
  The rate of live birth vs. still birth at delivery
Delivery mode | 6 weeks
  The mode of delivery (vaginal vs. cesarean vs. instrumental)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna General Hospital, Department of Obstetrics and Gynecology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farr A, Sustr V, Kiss H, Rosicky I, Graf A, Makristathis A, Foessleitner P, Petricevic L. Oral probiotics to reduce vaginal group B streptococcal colonization in late pregnancy. Sci Rep. 2020 Nov 12;10(1):19745. doi: 10.1038/s41598-020-76896-4. PMID 33184437